CLINICAL TRIAL: NCT00601354
Title: Comparing Orlistat/Alli to Orlistat/Alli Plus Guided Self-help Group Therapy in Overweight Binge Eaters
Brief Title: Adding Guided Self-Help Group Therapy to the Alli Weight Loss Program in Treating Binge Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Debra L. Safer, PI, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23MH066330 (NIH); K23MH066330 (NIH)
Record Dates: First submitted 2008-01-04; First posted 2008-01-28 (Estimated); Results first posted 2013-09-09 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-06

CONDITIONS: Overweight; Eating Disorders
Keywords: Binge Eating; Orlistat; Alli; Guided Self-Help
MeSH Terms: conditions — Overweight; Feeding and Eating Disorders; Bulimia | interventions — Orlistat

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emotion Regulation Group therapy + alli (Experimental): Group taking the weight loss medication orlistat (alli), in conjunction with the alli weight loss program, plus 12 weekly sessions of guided self-help group psychotherapy
  Interventions: Behavioral: Emotion regulation group therapy; Drug: Orlistat/alli program
- Orlistat/alli program meds only (Active Comparator): Group taking the weight loss medication orlistat (alli), in conjunction with the alli weight loss program alone
  Interventions: Drug: Orlistat/alli program

INTERVENTIONS:
Behavioral: Emotion regulation group therapy — Emotion regulation guided self-help group therapy involves twelve 2-hour sessions of guided self-help group psychotherapy.
  Other Names: emotion regulation guided self-help group therapy
  Arms: Emotion Regulation Group therapy + alli
Drug: Orlistat/alli program — The orlistat/alli program involves taking 60 mg orlistat three times a day and participating in the alli program, a comprehensive behavioral weight loss program with online access.
  Other Names: Alli

SUMMARY:
This study will evaluate the effectiveness of adding guided self-help group therapy to a weight loss program in achieving weight loss and reducing binge eating in overweight binge eaters.

DETAILED DESCRIPTION:
Binge eating disorder is one of the most common eating disorders, with more than 4 million Americans affected. Following a binge eating episode, in which a person eats an excessive amount of food in a short period of time, the person often experiences feelings of guilt, depression, embarrassment, and disgust. Beyond the emotional distress caused by binge eating, people who binge eat are at a higher risk for more serious health problems associated with weight gain. These health problems may include high blood pressure, diabetes, heart disease, high cholesterol, and certain types of cancer. Thus, seeking effective treatment for binge eating disorder is vital to an affected person's overall physical and mental well-being. Managed weight loss programs, combined with certain forms of psychotherapy, have shown success in providing the direction and proper motivation to eat healthily and to prevent future binge eating episodes. This study will evaluate the effectiveness of adding guided self-help group therapy to the alli weight loss program in achieving weight loss and reducing binge eating in overweight binge eaters.

Participation in this single-blind study will last 36 weeks. Initial assessments will be divided over two 1- to 2-hour sessions. These assessments will include a history of any medical illness, height and weight measurements, and an eating disorder evaluation. Participants will also answer several questionnaires about self-esteem, feelings of depression, and emotion and eating. Participants will then be randomly assigned to one of two treatment groups: the alli program with the use of the weight loss drug orlistat or the alli program with the use of orlistat plus guided self-help group psychotherapy. All participants will take the over-the-counter weight loss medication orlistat three times a day for 12 weeks in conjunction with the alli program, a comprehensive weight loss program with online access. Participants assigned to the psychotherapy group will also attend 12 weekly guided self-help group psychotherapy sessions. These sessions will include behavioral support for adapting to the lifestyle changes promoted by the alli weight loss program.

All participants will undergo 12 weeks of active participation, 18 weeks of maintenance, and 18 weeks of follow-up. At various intervals during the first 6 months of the study, participants will answer a short group of questions concerning current binge eating habits; adherence to prescribed food, activity, and medication plan; and emotional state. The initial assessments will be repeated at Weeks 12, 30, and 42.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index greater than 27
* Binge eating at least two times per week during the 6 months prior to study entry

Exclusion Criteria:

* Current psychosis
* Current suicidal ideations
* Pregnant
* Receiving concurrent psychotherapy
* Unstable on psychotropic medications for 3 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra L. Safer, MD, Principal Investigator — Stanford University Department of Psychiatry
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through newspaper advertisements and flyers. The study took place at an outpatient psychiatry department of a large university medical center.
Pre-assignment Details: There was no wash out, run-in, or transition following participant enrollment.Exclusion criteria are described previously. Main exclusion was weight less than 27 kg/m2.
Groups:
- OTC Orlistat + Guided Self-help Affect Regulation: Group taking the weight loss medication orlistat (alli), in conjunction with the alli weight loss program, plus 12 weekly sessions of guided self-help group psychotherapy
- OTC Orlistat /Medication Management Alone: Group taking the weight loss medication orlistat (alli), in conjunction with the alli weight loss program alone
Period: Overall Study
Arm/Group | OTC Orlistat + Guided Self-help Affect Regulation | OTC Orlistat /Medication Management Alone
Started | 8 | 9
Completed | 4 | 4
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OTC Orlistat + Guided Self-help Affect Regulation | OTC Orlistat /Medication Management Alone | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48.6 (11.2) | 50.1 (4.1) | 49.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: Change in weight in lbs from per to post treatment
Time Frame: 3 months: Measured from pre to post treatment
Population: Used intent-to-treat analysis
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | OTC Orlistat + Guided Self-help Affect Regulation | OTC Orlistat /Medication Management Alone
Number analyzed (Participants) | 8 | 9
lbs | 6.15 (14.36) | 3.61 (8.11)

2. Secondary Outcome: Binge Frequency
Description: frequency of objective binge days over prior 28 days
Time Frame: 3 months: Measured from pre to post treatment
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: % change objective binge days
Arm/Group | OTC Orlistat + Guided Self-help Affect Regulation | OTC Orlistat /Medication Management Alone
Number analyzed (Participants) | 8 | 9
% change objective binge days | 9.0 (2.13) | 12.11 (5.44)

3. Other Pre Specified Outcome: Weeks of Adherence to Orlistat
Time Frame: Number of adherent weeks over 1 year study
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: week of adherence to orlistat
Arm/Group | OTC Orlistat + Guided Self-help Affect Regulation | OTC Orlistat /Medication Management Alone
Number analyzed (Participants) | 8 | 9
week of adherence to orlistat | 13.8 (17.3) | 20.6 (19.1)

ADVERSE EVENTS:
Arm/Group | OTC Orlistat + Guided Self-help Affect Regulation | OTC Orlistat /Medication Management Alone
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No